CLINICAL TRIAL: NCT07288606
Title: Marginal Bone Loss in Implants Placed in Bone Level and Tissue Level
Brief Title: Analysising the Marginal Bone Loss, Torque and Implant Stability Placed in Bone and Tissue Level Dental Implants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, José López Lopez, Director, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022-033-1
Record Dates: First submitted 2024-06-12; First posted 2025-12-17 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Dental Implant; Implant Stability
Keywords: Bone level; tissue level; osseointegration; biomechanical analysis; implant design; Insertion torque

STUDY DESIGN:
Intervention Model Description: placement of dental implants in bone level and tissue level
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone Level (Experimental): Placement of a bone-level dental implant. The implant-abutment interface is at the level of the alveolar bone crest.
  Interventions: Procedure: Dental implant placement
- Tissue Level (Active Comparator): Placement of a tissue-level dental implant. The implant-abutment interface is located supracrestally, at the level of the soft tissue.
  Interventions: Procedure: Dental implant placement

INTERVENTIONS:
Procedure: Dental implant placement — Surgical placement of Bone-level and Tissue-level dental implants.

SUMMARY:
It is a prospective clinical study to compare two implants of the same brand of a similar design for implantation [either at the bone tissue level or at the soft tissue level], in order to evaluate the marginal bone loss of each dental implant in mm. 96 patients will be analyzed (an expected N of 48 per group, hoping to reach 100 implants per arm).

DETAILED DESCRIPTION:
it is a study to evualte the marginal bone loss in bone level and tissue level dental implants

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, over 18 years of age, who need dental implant placement for prosthetic rehabilitation. Whether partially or completely in both the maxilla and the mandible.
* Patients with residual alveolar ridge with at least 8 mm of bone height and 4 mm of width.
* Patients must have the ability to understand and decide when voluntarily signing the informed consent before carrying out any intervention related to the study.
* Patients who, after being informed about the objectives and procedures of the research, agree will sign the informed consent form. And they are ready to carry out the different study visits.

Exclusion Criteria:

* Patients with uncontrolled systemic diseases (ASA ≥ III).
* Patients who do not have 8mm bone height and/or 4mm width
* Patients who require bone regeneration
* Patients with severe periodontal disease or acute pericoronitis.
* Pregnant and breastfeeding women.
* Patients with Deficient or Inadequate Oral Hygiene.
* Patients with severe bruxism.
* Patients taking bisphosphonates or other antiresority medications.
* Smoker of more than 10 cigarettes/day.
* Patients with uncontrolled diabetes mellitus.
* Psychiatric illnesses or unrealistic expectations.
* Immunodepressed or immunocompromised patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Torque | up to 24 weeks
  N·cm
marginal bone loss | 6 months
  mm

CONTACTS AND LOCATIONS:
Overall Officials: JOSE L LOPEZ, MSC, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Odontologic, Barcelona, L'Hospitalet de Llobregat, Spain

DOCUMENTS (2):
  • Study Protocol (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT07288606/Prot_000.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT07288606/ICF_001.pdf